CLINICAL TRIAL: NCT00800124
Title: A Prospective Randomized Multicenter Study on Cemented and Non-cemented Hemiprosthesis in Older Patients With Dislocated Hip Fracture.
Brief Title: Study on Cemented Versus Non-cemented Hemiarthroplasty in Elderly With Hip Fractures
Acronym: CNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Rikshospitalet University Hospital (Other); Sykehuset Buskerud HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNC2008
Record Dates: First submitted 2008-11-27; First posted 2008-12-01 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Hip Fracture
Keywords: hip fracture; hemiprosthesis; bone cement; clinical outcome
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Cemented hemiprosthesis
- 2 (Active Comparator): Non-cemented hemiprosthesis
  Interventions: Procedure: cemented Landos prosthesis vs. uncemented Landos prosthesis

INTERVENTIONS:
Procedure: cemented Landos prosthesis vs. uncemented Landos prosthesis — randomization between the cemented and non-cemented prosthesis.
  Other Names: Titanium prosthesis; Corail uncemented prosthesis
  Arms: 2

SUMMARY:
The objective is to study the overall frequency and cumulative rate (during one year) of clinical morbidity (defined as any hospitalization without fatal outcome) and mortality in all consecutive patients undergoing HF surgery (pins and prosthetic implants) and compare this to the group of patients receiving prosthetic implants and further find out if there is a difference between the non-cemented and cemented groups.

Between the same prosthetic groups, the investigators want to study the overall frequency of in-hospital subclinical organ damage and dysfunction of myocardium, liver and lungs, using biochemical plasma markers. Finally, the investigators want to perform perioperative cost benefit calculations and out of hospital quality of life analysis between the surgical groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Garden 3 or 4 fracture in acute hip fractures.
* Age over 75 years.

Exclusion Criteria:

* Patient or relative refuse enrollment

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 334 (Actual)
Dates: Start 2005-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ove Talsnes, MD, Principal Investigator — Sykehsuet Innlandet, Elverum
Locations (1):
- Sykehuset Innlandet, Elverum, Elverum, Hedmark, Norway